CLINICAL TRIAL: NCT03618849
Title: Safety and Feasibility of Transcranial Direct Current Stimulation in Pediatric Acquired Brain Injury (tDCS in Pediatric ABI)
Brief Title: tDCS in Pediatric Acquired Brain Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: limited recruitment
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00174966
Record Dates: First submitted 2018-06-13; First posted 2018-08-07 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Acquired Brain Injury; Disorders of Consciousness
Keywords: Acquired Brain Injury; Transcranial Direct Current Stimulation; Pediatric; Safety; Feasibility
MeSH Terms: conditions — Brain Injuries; Consciousness Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Dosage-escalation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham tDCS (Experimental): Post initial screening and baseline data collection, all study participants (a single cohort of patients) will receive a single dose of sham tDCS for 20 minutes over the left dorsolateral prefrontal cortex (DLPFC) or the primary motor cortex in conjunction with Mozart piano sonata. For sham tDCS, the current will be ramped up and immediately ramped down for 30 seconds. The sham tDCS session will be preceded and followed by behavioral assessments.
  Interventions: Device: tDCS
- 1-mA tDCS (Experimental): Post sham-tDCS, we will determine the eligibility of the participant to receive 1 mA of real tDCS based on the occurrence of adverse events and seizures occurring within 5 days of the sham session. After a minimum of 5 days post-sham stimulation (and typically around 7 days later), the participant will receive a single dose of 1-mA current (for head circumference >52 cm; children with head circumference 43-52cm will receive 0.5-mA) over left DLPFC or M1 in conjunction with Mozart piano sonata. The participant will receive 1-mA current for 20 minutes; the current will be ramped up for 30 seconds, will held constant at the determined intensity for 20 minutes, and then ramped down for 10 seconds. The 1-mA tDCS session will be preceded and followed by behavioral assessments.
  Interventions: Device: tDCS
- 2-mA tDCS (Experimental): Post 1-mA tDCS, we will again determine the eligibility of the participant to receive 2 mA current. After a minimum of 5 days post-1 mA stimulation (typically 7 days), the participant will receive a single dose of 2-mA current (if head circumference >52cm; children with head circumference 43-52cm will receive 1-mA) over left DLPFC or M1 in conjunction with Mozart piano sonata. The participant will receive 2-mA current for 20 minutes; the current will be ramped up for 30 seconds, will held constant at the determined intensity for 20 minutes, and then ramped down for 10 seconds. The 2-mA tDCS session will be preceded and followed by behavioral assessments.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Real and sham tDCS/Mozart piano sonata (K.448)
  Other Names: transcranial direct current stimulation; non-invasive brain stimulation

SUMMARY:
In this preliminary study, we will examine the safety, tolerability, and feasibility of transcranial direct current stimulation (tDCS), in the setting of dosage escalation, as a candidate intervention for children with Acquired Brain Injury (ABI).

DETAILED DESCRIPTION:
Previous studies have demonstrated that transcranial direct current stimulation (tDCS) is safe and effective in adults with chronic Acquired Brain Injury. Limited data have established the safety of tDCS in children with neuropsychiatric and neuromotor disorders. However, these tDCS safety paradigms may not be relevant to children with ABI due to their abnormal brain structure and function, decreased ability to communicate, variable symptomology, and time-consuming care needs that exist in this population.

In this open-label, single-group, dosage escalation study, investigators aim to assess the safety, tolerability, and feasibility of incrementally higher tDCS currents in 10 pediatric patients with ABI on an inpatient rehabilitation unit. The study will include up to three sessions of tDCS (sham, 1mA, and then 2 mA) either over the left dorsolateral prefrontal cortex or over the primary motor cortex based on the goal to evaluate change in either cognitive or motor function. We will also explore whether tDCS improves consciousness in pediatric DOC. Mozart classical music, as a concurrent intervention, will be played during sham, 1 mA, and 2 mA tDCS applications.

ELIGIBILITY:
Inclusion Criteria:

* Age 5 through 17 years
* History of acquired brain injury.
* Currently inpatient at the Kennedy Krieger Rehabilitation Unit.
* Parent and child proficient in English.

Exclusion Criteria:

* Patients with extensive focal lesions in the left dorsolateral prefrontal cortex (DLPFC) and bilateral primary motor cortex as determined by review of imaging and/or imaging reports obtained as part of clinical care.
* Youth with known seizures in the month prior to study enrollment.
* Participants with non-convulsive seizures and/or interictal epileptiform discharges observed on study screening extended EEG.
* Females with confirmed pregnancy on urine test.
* Youth with history of craniotomy surgery, metallic cerebral, cochlear or electronic implant in the head or neck area, or ventricular shunt or pacemaker.
* Patients requiring daytime mechanical ventilation.
* Children with head circumference less than 43 cm
* Bilateral severe or profound hearing loss
* Presence of hairstyle interfering with tDCS application and/or high quality EEG signal
* Youth in foster care.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in adverse events (skin problems and/or seizures) as a measure of safety | Baseline (1-7 days), post-stimulation (within 30-minutes), follow-up (24 hours, 48 hours, 5 days)
  Adverse Event Form Questionnaire: Assessment of change from baseline and post-sham stimulation to post- stimulation (1 mA, 2 mA) and follow-up using a detailed assessment of participant's symptoms (skin problems and/or seizures) as related to transcranial direct current stimulation (tDCS) intervention.
Changes in pain and discomfort as a measure of safety and tolerability | Baseline (1-7 days), pre-during-post stimulation (pre-stimulation: within 30 minutes, during: within 20 minutes, post-stimulation: within 30-minutes)
  Face, Legs, Activity, Cry and Consolability Scale (FLACC) Questionnaire: Assessment of change from baseline and post-sham stimulation to pre-during-post stimulation (1 mA, 2 mA) using an observation tool that will measure pain and discomfort as related to transcranial direct current stimulation (tDCS) in children with decreased communication and cognitive impairment.
Disruption of Care Form | Up to 26 Days
  Questionnaire: Assessment of interruption of inpatient care due to child's participation in the study.
Family Feedback Form | 5 days after the end of the last stimulation session.
  Questionnaire: Assessment to receive feedback about the satisfaction in the study from the parent/guardian/caregiver of the participant.
Number of participants with adverse events as related to tDCS | Up to 26 Days
  The information on number of participants with adverse events will be collected from the beginning of sham tDCS until the end of the last tDCS session.

SECONDARY OUTCOMES:
Changes in Neurobehavioral functioning | Up to 4 months
  Modified Functional Reach Task, Grooved Pegboard, Digit Span, or Coma-Recovery Scale Revised: Task chosen based on child's functional status and assessment of change from baseline, post-sham stimulation, and pre-stimulations (1 mA, 2 mA).

CONTACTS AND LOCATIONS:
Overall Officials: Stacy J Suskauer, MD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thibaut A, Di Perri C, Chatelle C, Bruno MA, Bahri MA, Wannez S, Piarulli A, Bernard C, Martial C, Heine L, Hustinx R, Laureys S. Clinical Response to tDCS Depends on Residual Brain Metabolism and Grey Matter Integrity in Patients With Minimally Conscious State. Brain Stimul. 2015 Nov-Dec;8(6):1116-23. doi: 10.1016/j.brs.2015.07.024. Epub 2015 Sep 14. PMID 26471400
- [Background] Krishnan C, Santos L, Peterson MD, Ehinger M. Safety of noninvasive brain stimulation in children and adolescents. Brain Stimul. 2015 Jan-Feb;8(1):76-87. doi: 10.1016/j.brs.2014.10.012. Epub 2014 Oct 28. PMID 25499471
- [Background] Rivera-Urbina GN, Nitsche MA, Vicario CM, Molero-Chamizo A. Applications of transcranial direct current stimulation in children and pediatrics. Rev Neurosci. 2017 Feb 1;28(2):173-184. doi: 10.1515/revneuro-2016-0045. PMID 27997354
- [Background] Gillick BT, Feyma T, Menk J, Usset M, Vaith A, Wood TJ, Worthington R, Krach LE. Safety and feasibility of transcranial direct current stimulation in pediatric hemiparesis: randomized controlled preliminary study. Phys Ther. 2015 Mar;95(3):337-49. doi: 10.2522/ptj.20130565. Epub 2014 Nov 20. PMID 25413621
- [Background] Giustini A, Pistarini C, Pisoni C. Traumatic and nontraumatic brain injury. Handb Clin Neurol. 2013;110:401-9. doi: 10.1016/B978-0-444-52901-5.00034-4. PMID 23312659
- [Background] Ashwal S. Medical aspects of the minimally conscious state in children. Brain Dev. 2003 Dec;25(8):535-45. doi: 10.1016/s0387-7604(03)00095-0. PMID 14580666
- [Background] Giacino JT, Trott CT. Rehabilitative management of patients with disorders of consciousness: grand rounds. J Head Trauma Rehabil. 2004 May-Jun;19(3):254-65. doi: 10.1097/00001199-200405000-00006. PMID 15247847
- [Background] Ragazzoni A, Cincotta M, Giovannelli F, Cruse D, Young GB, Miniussi C, Rossi S. Clinical neurophysiology of prolonged disorders of consciousness: From diagnostic stimulation to therapeutic neuromodulation. Clin Neurophysiol. 2017 Sep;128(9):1629-1646. doi: 10.1016/j.clinph.2017.06.037. Epub 2017 Jun 29. PMID 28728060
- [Background] Chung MG, Lo WD. Noninvasive brain stimulation: the potential for use in the rehabilitation of pediatric acquired brain injury. Arch Phys Med Rehabil. 2015 Apr;96(4 Suppl):S129-37. doi: 10.1016/j.apmr.2014.10.013. Epub 2014 Nov 6. PMID 25448248
- [Derived] Saleem GT, Ewen JB, Crasta JE, Slomine BS, Cantarero GL, Suskauer SJ. Single-arm, open-label, dose escalation phase I study to evaluate the safety and feasibility of transcranial direct current stimulation with electroencephalography biomarkers in paediatric disorders of consciousness: a study protocol. BMJ Open. 2019 Aug 10;9(8):e029967. doi: 10.1136/bmjopen-2019-029967. PMID 31401607